CLINICAL TRIAL: NCT03297385
Title: Dynamics of Androgen Receptor Genomics and Transcriptomics After Neoadjuvant Androgen Ablation
Acronym: DARANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N14DAR
Record Dates: First submitted 2017-04-13; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer; DNA; Androgen Receptor Abnormal
Keywords: Prostate Cancer; Androgen Receptor Genomics; Enzalutamide; Prostatectomy; Neoadjuvant androgen ablation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: A phase II prospective single-arm analysis. With a power of 80% to detect an expected reduction in positive surgical margin rate from 34% to 17% we will have to included 55 men. For the AR/DNA interaction patients will serve as there own control since biopsies will be taken before and after enzalutamide treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostatectomy after enzalutamide (Experimental): This is a single-arm study. Patients will have biopsies, after which they will receive enzalutamide for 3 months.
  After 3 months they will have a prostatectomy.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Men with localized prostate cancer will undergo an additional set of targeted tumor biopsies and will be subsequently treated with 3 months of enzalutamide. The prostatectomy specimen will be additionally sampled, ex vivo.
  Other Names: Xtandi

SUMMARY:
Rationale: Understanding the mechanisms of enzalutamide as an androgen receptor inhibitor in early prostate cancer could lead to improved patient selection for treatment.

Objective: To study the effects of enzalutamide on surgical margin status and AR / DNA interaction and gene expression.

Intervention : Men with localized prostate cancer will undergo an additional set of targeted tumor biopsies and will be subsequently treated with 3 months of enzalutamide. The prostatectomy specimen will be additionally sampled, ex vivo.

DETAILED DESCRIPTION:
Rationale: Understanding the mechanisms of enzalutamide as an androgen receptor inhibitor in early prostate cancer could lead to improved patient selection for treatment.

Objective: To study the effects of enzalutamide on surgical margin status and AR / DNA interaction and gene expression.

Study design: A phase II prospective single-arm analysis. With a power of 80% to detect an expected reduction in positive surgical margin rate from 34% to 17% the investigators will have to included 55 men. For the AR/DNA interaction patients will serve as there own control since biopsies will be taken before and after enzalutamide treatment.

Study population: Patients over 18 years of age with localized prostate cancer that are planned for prostatectomy.

Intervention : Men with localized prostate cancer will undergo an additional set of targeted tumor biopsies and will be subsequently treated with 3 months of enzalutamide. The prostatectomy specimen will be additionally sampled, ex vivo.

Main study parameters/endpoints: 1. The effects of neoadjuvant androgen ablation on tumor downstaging. 2. The genetic and transcriptional changes caused by neoadjuvant androgen ablation by enzalutamide.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Burden and risks: Patients will be submitted to an additional set of 4 tumor targeted biopsies under local anesthesia and antibiotic prophylaxis. This comprises a 5 minute intervention with an elevated (2%) risk of postbiopsy urinary tract infection. Additionally oral enzalutamide treatment for a period of 3 months will result in temporary signs of androgen ablation such as: hot flushes (20%), headache (12%), diarrhea (1%), and seizures (0.9%). Benefits: neoadjuvant enzalutamide treatment has been shown to result in tumor and prostate downsizing. Earlier neoadjuvant androgen ablation studies with other agents have shown a reduced positive surgical margin rate and reduced intraoperative blood loss

ELIGIBILITY:
Inclusion Criteria:

1. Men over 18 years of age.
2. clinically non-metastasized prostate cancer, tumor that can be imaged (TRUS or MRI) in order to allow for accurate preoperative biopsies.
3. Gleason score 7-10
4. written informed consent
5. WHO performance 0-1

Exclusion Criteria:

1. A history of seizures.
2. Clinically nodal metastases.
3. Prostatitis or urinary tract infection.
4. Androgen ablative therapy within 6 weeks of inclusion (including 5 alpha-reductase inhibitors).
5. Tumor of the prostate that can not be visualized by TRUS or MRI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Effects of enzalutamide on tumor downstaging | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  To study the effects of enzalutamide on surgical margin status and AR / DNA interaction and gene expression.
Genetic and transcriptional changes caused by enzalutamide | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  The genetic and transcriptional changes caused by neoadjuvant androgen ablation by enzalutamide.

SECONDARY OUTCOMES:
Clinical down-staging of enzalutamide pretreatment | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  To assess the effects of 3 months enzalutamide pretreatment on clinical down-staging
AR-chromatin binding alterations and Ki-67 expression | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  Study the correlation between AR-chromatin binding alterations and Ki-67 expression.
AR-dependant genes such as PSA, human kallikrein and PSMA | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  Compare the AR-chromatin binding with expression alterations of known AR-dependent genes such as PSA, human kallikrein and PSMA.
Gleason grading | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  Compare AR-chromatin binding patterns with Gleason grading.
Find associated genes in prostate tissue, using tissue microarray (TMA). | From baseline (prior to treatment), until disease progression or as long as treatment is tolerated or until study completion (60 months).
  Find associated genes on TMA derived from prostatectomy specimens.

REFERENCES:
- [Derived] Zhang M, Moreno-Rodriguez T, Quigley DA. Why ARNT Prostate Tumors Responding to Enzalutamide? Cancer Discov. 2022 Sep 2;12(9):2017-2019. doi: 10.1158/2159-8290.CD-22-0702. PMID 36052502